CLINICAL TRIAL: NCT06953115
Title: Vagal Autonomic Stimulation Physiotherapy (With Trigger Point Release) as an Adjunct to Personalized Antihypertensive Management of Gestational Hypertension Syndrome and Preeclampsia
Brief Title: Vagal Stimulation Therapy and Preeclampsia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Internacional René Mey (Other)
Collaborators: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Carlos Alberto Garcia Becerra, Principal Investigator, Fundación Internacional René Mey, Fundación Internacional René Mey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2025-785-018
Record Dates: First submitted 2025-04-03; First posted 2025-05-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Gestational Hypertension; Preeclampsia
Keywords: Hypertension, Pregnancy-Induced; Gestational Hypertension; Pre-Eclampsia; Preeclampsia; Physical Therapy Techniques; Modalities, Physical Therapy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Clinical trial with an open-label intervention administration
Who Masked: Participant, Investigator
Masking Description: The study is designed as a double-blind, non-pharmacological clinical trial with a pre-test/post-test design. Both the participants and the outcome evaluator conducting the statistical analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagal Stimulation Physiotherapy with Trigger Point Release (TEV Group). (Experimental): Administration of physiotherapy sessions for vagal stimulation with trigger point release, in addition to personalized antihypertensive treatment.
  Interventions: Other: Vagal stimulation physiotherapy with trigger point release
- Positional Release Therapy (TLP Group). (Active Comparator): Administration of positional release therapy sessions, in addition to personalized antihypertensive treatment.
  Interventions: Other: Positional Release Therapy

INTERVENTIONS:
Other: Vagal stimulation physiotherapy with trigger point release — The patient will be instructed to remain in a seated position, with the knee slightly ahead of the feet and the feet firmly planted on the floor, with the hips higher than the knees. The therapist will stand behind the patient. Myofascial release will be performed on the upper trapezius (UT) while the patient slowly turns their head from side to side and lets it drop forward. The therapist will then apply pressure on the opposite side of the rotation.
  * Therapist's position: Behind the patient.
  * Patient's position: Seated with the spine in a neutral position.
  Arms: Vagal Stimulation Physiotherapy with Trigger Point Release (TEV Group).
Other: Positional Release Therapy — A 30-minute session of positional release therapy will be provided every two weeks, in addition to personalized antihypertensive treatment, from the start of treatment (T0) until the final measurement (days 28 to 35 after obstetric resolution).
  Keeping the cervical spine in a neutral position, the participant will be asked to lie down in a relaxed supine position. The therapist will progressively apply more pressure to the trigger points identified with their thumb. In the next step, the therapist will move to a more comfortable position that exerts less stress. The therapist will passively hold the patient's upper limbs in an abducted position, with a rest period between each repetition.
  * Therapist's position: On the side of the patient.
  * Patient's position: Supine.
  Arms: Positional Release Therapy (TLP Group).

SUMMARY:
Preeclampsia is one of the most common and serious complications of pregnancy, affecting both the mother and baby. It is a condition characterized by high blood pressure and can lead to severe complications, including neurological issues and reduced blood flow to the placenta. Preeclampsia is responsible for a significant number of maternal and perinatal deaths worldwide, with an estimated 14% of maternal mortality in Mexico linked to this condition.

Recent research suggests that disruptions in the body's autonomic nervous system, specifically the balance between the sympathetic and parasympathetic systems, play a role in the development of preeclampsia. The vagus nerve, which is part of the parasympathetic system, has been shown to regulate inflammation and blood pressure. Stimulating this nerve through pharmacological, magnetic, electrical, or physical therapy techniques has shown promise in preclinical models for improving blood pressure control and reducing complications associated with preeclampsia.

Trigger point release therapy modulates the nervous system by reducing sympathetic activity, promoting blood vessel relaxation, lowering heart rate, and enhancing circulation. When combined with standard antihypertensive treatment, this approach may offer additional benefits for blood pressure regulation.

This study aims to evaluate the effects of vagal autonomic stimulation physiotherapy using trigger point release therapy as a complementary treatment for pregnant women with preeclampsia. Participants will be randomly assigned to receive either standard antihypertensive treatment with positional release therapy (control group) or the same treatment combined with vagal stimulation physiotherapy (intervention group). Researchers will assess the intervention's effectiveness in controlling blood pressure and improving overall maternal and fetal health outcomes.

By investigating this non-invasive, drug-free approach, this study aims to offer new strategies for managing preeclampsia, potentially improving maternal and fetal health while reducing reliance on medication.

DETAILED DESCRIPTION:
Among hypertensive disorders of pregnancy, preeclampsia is the most common medical complication and is associated with high medical and social costs, making it a significant public health concern.

Although its global prevalence is unknown, preeclampsia is implicated in 14% of maternal deaths worldwide. In Mexico, it accounts for approximately 14% of maternal mortality, corresponding to a rate of 30.4 per 100,000 live births, and 17.2% of total perinatal deaths. Of these maternal deaths, 30% to 70% result from neurological complications where cerebral autoregulation is lost, leading to vasospasm, reduced blood flow, and ischemic and infarcted areas in the placenta.

Recent evidence suggests that dysregulation of the cholinergic anti-inflammatory pathway (CAP) may contribute to preeclampsia development. This pathway connects the central nervous system-via the vagus nerve-to mechanisms regulating inflammation in the body. It is influenced by the downregulation of the α7 nicotinic acetylcholine receptor, which has been associated with systemic inflammation in preeclampsia. Additionally, some electrical, pharmacological, magnetic, and physical vagal stimulation techniques targeting this pathway have shown promising results in preclinical models of preeclampsia, making vagus nerve activation a potential strategy for managing this pregnancy complication. Clinically, various vagal stimulation techniques, such as deep breathing, progressive relaxation, and transcranial magnetic stimulation, have been approved for treating depression and epilepsy in pregnant women.

Primarily linked to the parasympathetic nervous system, the vagus nerve is also influenced by the sympathetic nervous system through peripheral receptors. Trigger point stimulation therapy in physiotherapy can block sympathetic nervous system activity, reducing peripheral vascular resistance, venous return, heart rate, and myocardial contractility by promoting systemic arterial and venous vasodilation. In this context, physiotherapy involving trigger point release could serve as an adjunct treatment for blood pressure control in preeclamptic patients by modulating the peripheral nervous system. However, its impact on autonomic tone has not yet been reported.

This study aims to explore the benefits of vagal stimulation through trigger point release, combined with medical treatment for preeclampsia-an approach that has not been fully investigated in our setting. This protocol presents a non-invasive complementary technique to support personalized pharmacological management of preeclamptic patients. By enhancing the vasorelaxant response derived from autonomic nervous system activity, this intervention may help reduce blood pressure levels and biochemical markers associated with preeclampsia.

Objective: To determine the effect of vagal autonomic stimulation physiotherapy with trigger point release on hemodynamic control compared to positional release therapy as adjuvant treatments in personalized antihypertensive therapy for gestational hypertension syndrome preeclampsia.

Methods: This is an Experimental, randomized, double-blind, parallel-group clinical trial with an open-label intervention administration, with a control group (2:1 ratio), designed to assess the effectiveness of vagal stimulation physiotherapy with trigger point release as an adjuvant treatment for mild preeclampsia in pregnant women. The study will be conducted over 12 months at several hospitals of the Mexican Institute of Social Security.

Participants:

Women over 18, beneficiaries of the Mexican Institute of Social Security (IMSS), diagnosed with mild preeclampsia, will be randomly assigned to one of two groups:

1. Intervention group: Receives vagal stimulation physiotherapy with trigger point release every two weeks, along with personalized antihypertensive treatment.
2. Control group: Receives positional release therapy every two weeks, along with personalized antihypertensive treatment.

Study Design:

* Blinding: Double-blind (patients and researcher performing statistical analysis).
* Sample Size: 210 patients (147 in the experimental group, 63 in the control group).
* Randomization: Block randomization generated by computer.

Inclusion Criteria: Outpatient pregnant women aged 18 years or older who are attending their first obstetrics consultation at the Regional General Hospitals of IMSS Jalisco with a confirmed diagnosis of mild preeclampsia. Participants must have no prior antihypertensive treatment and must be willing to participate by signing an informed consent form.

Exclusion Criteria: Patients with chronic hypertension, concomitant organ dysfunction, or immunological diseases will be excluded from the study. Additionally, those with severe preeclampsia or any chronic condition complicating pregnancy will not be eligible. Patients diagnosed with gestational trophoblastic disease requiring uterine evacuation or choriocarcinoma will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient female patients over 18 years old, attending their first appointment and seen in the obstetrics outpatient clinic at the Regional General Hospitals of IMSS Jalisco, with a pregnancy complicated by confirmed mild preeclampsia.
* No prior treatment.
* Willing to participate by signing an informed consent form.

Exclusion Criteria:

* Patients with chronic hypertension.
* Concomitant organ dysfunction.
* Immunological diseases.
* Patients with severe preeclampsia or chronic conditions concomitant with pregnancy.
* Patients with gestational trophoblastic disease requiring uterine evacuation or choriocarcinoma associated with hypertension.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in participants' blood pressure from baseline (T0), every 2 weeks (T1, T2, T3...), until the end of the evaluation period (TX). | From baseline until weeks 4 to 5 after obstetric resolution.
  Observed changes in the measurement of participants' diastolic and systolic blood pressure, recorded at baseline (T0), every 2 weeks (T1, T2, T3...), until the end of the evaluation period (TX).
Changes in participants' heart rate from baseline (T0), every 2 weeks (T1, T2, T3...), until the end of the evaluation period (TX). | From baseline until weeks 4 to 5 after obstetric resolution.
  Observed changes in the measurement of participants' heart rate, recorded at baseline (T0), every 2 weeks (T1, T2, T3...), until the end of the evaluation period (TX).

SECONDARY OUTCOMES:
Biochemical parameters of renal function (Changes in serum creatinine levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum creatinine levels in the participants, measured in milligrams per milliliter (mg/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of renal function (Changes in serum Urea levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum Urea levels in the participants, measured in milligrams per milliliter (mg/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of renal function (Changes in serum uric acid levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum uric acid levels in the participants, measured in milligrams per milliliter (mg/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of renal function (Changes in Glomerular filtration rate in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in Glomerular filtration rate in the participants, measured in milliliters per minute per 1.73 square meters of body surface area (mL/min/1.73), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Hematological parameters (Changes in complete blood count with platelet count in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in complete blood count with platelet count in the participants, measured in cells per cubic millimeter (cel/mm3), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum aspartate aminotransferase levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum aspartate aminotransferase levels in the participants, measured in milli-international units per milliliter (mUI/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum alanine aminotransferase levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum alanine aminotransferase levels in the participants, measured in milli-international units per milliliter (mUI/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum lactate dehydrogenase levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum lactate dehydrogenase levels in the participants, measured in milli-international units per milliliter (mUI/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum gamma-glutamyl transferase levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum gamma-glutamyl transferase levels in the participants, measured in milli-international units per milliliter (mUI/mL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum total protein levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum total protein levels in the participants, measured in grams per deciliter (g/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum albumin levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum albumin levels in the participants, measured in grams per deciliter (g/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum globulin levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum globulin levels in the participants, measured in grams per deciliter (g/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum albumin/globulin ratio in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum albumin/globulin ratio in the participants, from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum total cholesterol levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum total cholesterol levels in the participants, measured in milligrams per deciliter (mg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum HDL cholesterol levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum HDL cholesterol levels in the participants, measured in milligrams per deciliter (mg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum LDL cholesterol levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum LDL cholesterol levels in the participants, measured in milligrams per deciliter (mg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum VLDL cholesterol levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum VLDL cholesterol levels in the participants, measured in milligrams per deciliter (mg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical parameters of hepatic function (Changes in serum triglyceride levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum triglyceride levels in the participants, measured in milligrams per deciliter (mg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical Parameters of Inflammatory and Endothelial Dysfunction Response (Changes in serum C-reactive protein levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum C-reactive protein levels in the participants, measured in milligrams per deciliter (mg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical Parameters of Inflammatory and Endothelial Dysfunction Response (Changes in serum D-dimer levels in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in serum D-dimer levels in the participants, measured in micrograms per deciliter (μg/dL), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical Parameters of Inflammatory and Endothelial Dysfunction Response (Changes in prothrombin time in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in prothrombin time in the participants, measured in seconds (seg), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).
Biochemical Parameters of Inflammatory and Endothelial Dysfunction Response (Changes in activated partial thromboplastin time in the participants) | From baseline until 4 to 5 weeks after obstetric resolution.
  Changes in activated partial thromboplastin time in the participants, measured in seconds (seg), from baseline (T0) and every 2 weeks thereafter (T1, T2, T3...) until the end of the evaluation period (TX).

CONTACTS AND LOCATIONS:
Overall Officials: Luz Ma. Adriana Balderas-Peña, Ph.D., Study Chair — Unidad de Investigación Biomédica 02, UMAE HE CMNO IMSS; René Jaques Mey, Dr. h.c., Principal Investigator — Fundación Internacional René Mey; Juliette Myriam Laure, M.Sc., Principal Investigator — Fundación Internacional René Mey; Carlos A. García-Becerra, M.Sc., Principal Investigator — Fundación Internacional René Mey
Locations (4):
- Mexico (4):
  - Unidad de Investigación Biomédica 02, UMAE HE CMNO IMSS, Guadalajara, Jalisco
  - Hospital General de Zona 110, IMSS, Guadalajara, Jalisco
  - Hospital General de Zona 46, IMSS, Guadalajara, Jalisco
  - Hospital General de Zona 180, IMSS, Tlajomulco de Zúñiga, Jalisco

IPD SHARING:
Plan to Share IPD: Undecided